CLINICAL TRIAL: NCT05255523
Title: A Single Arm，Multicenter，Real-world Observational Study of Pyrotinib Plus Trastuzumab After First-line TH (P) Treatment With HER-2 Positive Breast Cancer
Brief Title: Pyrotinib Plus Trastuzumab After First-line TH (P) Treatment With HER-2 Positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Advanced Breast Cancer
Keywords: pyrotinib;CNS;breast cancer; HER-2 positivity
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Pyrotinib：400mg qd po continuous medication Capecitabine: 1000 mg/m2 bid po for 14 consecutive days with 7 days off, every 21 days as a cycle.
  Interventions: Drug: pyrotinib

INTERVENTIONS:
Drug: pyrotinib — After 4-6 cycles of taxane chemotherapeutics combined with trastuzumab±pertuzumab, the assessment result reaches CR or PR, and the subsequent sequential pyrrotinib plus capecitabine±trastuzumab to CNS Progress
  Other Names: capecitabine

SUMMARY:
The purpose of this study is to assess the effect of pyrotinib

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of pyrotinib combined with trastuzumab in the maintenance phase delay/reduction of brain metastases after first-line TH(P) therapy for HER-2-positive advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years old, female;
2. HER2 positive advanced breast cancer diagnosed by pathology, cytology or radiology, including inoperable breast cancer with stage IV, or recurrent/metastatic breast cancer.HER-2 positivity was confirmed by histopathological test: immunohistochemistry(IHC) results of 3 + or in situ hybridization (ISH) results of amplification of HER2;
3. Disease progression occurs after treatment with trastuzumab (stopping the drug for more than 12 months) or newly diagnosed IV stage breast cancer patients;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
5. Life expectancy greater than or equal to 6 months;
6. The main organs function well, and the inspection indicators meet the following requirements:

1) For results of blood routine test HB≥90g/L; ANC≥1.5×109/L; PLT≥90×109/L; 2) For results of blood biochemical test ALT and AST≤2×ULN, but≤5×ULN if the transferanse elevation is due to liver metastases； TBIL≤1.5×ULN； Serum creatinine ≤1.5×ULN; 7. The researchers believed that the subjects were preference to benefit; 8. Participants were willing to join in this study, and written informed consent.

Exclusion Criteria:

1. Patients with brain metastases by CT or MRI;
2. More factors affecting of oral drugs (gastrointestinal surgery history, inability to swallow, chronic diarrhea, intestinal obstruction);
3. Study drug and excipient allergy;
4. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
5. Pregnant or lactating female patients;
6. Less than 4 weeks from the last clinical trial;
7. The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-11-05 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of first progression with brain metastases | 24 month
  Incidence of first progression with brain metastases

SECONDARY OUTCOMES:
ORR without CNS | 24 month
  Baseline to measured stable disease without central nervous system
TTBM | 24 month
  Time to brain metastases

IPD SHARING:
Plan to Share IPD: No